CLINICAL TRIAL: NCT02031016
Title: A Randomised Clinical Trial Evaluating the Effect of Remifentanil vs Fentanyl During Cardiac Surgery on the Incidence of Chronic Thoracic Pain
Brief Title: Remifentanil vs Fentanyl During Cardiac Surgery and Chronic Thoracic Pain
Acronym: REFLECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Catherijne Knibbe, Prof. Dr., St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REFLECT study
Record Dates: First submitted 2013-12-16; First posted 2014-01-09 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Pain; Sternotomy; Remifentanil; Fentanyl
Keywords: Chronic thoracic pain; Remifentanil; Fentanyl; sternotomy
MeSH Terms: conditions — Chronic Pain | interventions — Fentanyl; Remifentanil

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Fentanyl (Active Comparator): fentanyl bolus injections on an "as needed" base, next to the fentanyl bolus injections on predetermined times; before incision, at sternotomy, at aorta canulation and at opening of the pericardium.
  Interventions: Drug: Fentanyl
- Remifentanil (Active Comparator): remifentanil, starting with 0.15 ug/Ideal Body Weight(IBW)(kg)/min, next to fentanyl bolus injections (200-500 ug) on predetermined times; before incision, at sternotomy, at aorta canulation and at opening of the pericardium.
  Interventions: Drug: Remifentanil; Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — fentanyl bolus injections on an "as needed" base, NEXT TO the fentanyl bolus injections on predetermined times; before incision, at sternotomy, at aorta canulation and at opening of the pericardium.
  Other Names: Sublimaze
  Arms: Fentanyl
Drug: Remifentanil — starting with 0.15 ug/IBW(kg)/min, next to fentanyl bolus injections (200-500 ug) on predetermined times; before incision, at sternotomy, at aorta canulation and at opening of the pericardium.
  Other Names: Ultiva
  Arms: Remifentanil
Drug: Fentanyl — fentanyl bolus injections on predetermined times; before incision, at sternotomy, at aorta canulation and at opening of the pericardium.
  Other Names: Sublimaze

SUMMARY:
This study will investigate the influence of intra-operative use of remifentanil versus fentanyl on the percentage of patients with chronic thoracic after cardiac surgery via sternotomy. Secondary quantitative sensory testing is performed to determine thermal and electrical detection and pain threshold and the difference in pain variability scoring. Postoperative pain scores, analgesic use, genetic variances and costs are measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery via sternotomy (Coronary artery bypass graft (CABG) and/or valve replacement)
* Patients admitted to the ICU or PACU in the St. Antonius hospital
* Patients between 18 and 85 years old
* Patients weighing between 45 and 140 kg
* Written informed consent

Exclusion Criteria:

* Pregnancy/ breastfeeding
* Language barrier
* History of drug abuse
* Neurologic condition such as peripheral neuropathy
* Known remifentanil, fentanyl, morphine or paracetamol allergy
* Body Mass Index (BMI) > 35 kg/m2
* Prior cardiac surgery (re-operations);
* Patients with chronic pain conditions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Chronic thoracic pain | 1 year
  The percentage of patients reporting chronic thoracic pain one year after cardiac surgery.

SECONDARY OUTCOMES:
Chronic thoracic pain | 3 and 6 months
  The percentage of patients reporting chronic thoracic pain three months and six months after cardiac surgery
Mean Numerical Rating Scale (NRS) score | 3, 6 and 12 months
  The mean NRS score of patients with chronic thoracic pain three months and six months after cardiac surgery.
Quality of life | 3, 6 and 12 months
  The quality of life (QoL) three months, six months and one year after surgery.
Thermal detection and pain thresholds | preoperative, 3 days postoperative and 1 year after surgery
  The difference in postoperative pain thresholds three days and one year after cardiac surgery compared to the preoperative pain threshold (baseline)
Pain variability | preoperative, 3 days and 1 year postoperative
  Pain variability measured with a paradigm with electrical stimuli in only a part of the participants. The difference in pain variability preoperative, three days postoperative and one year after cardiac surgery.
Use of analgesics during and after hospitalization | 3 days during hospitalization and 3,6,12 months post surgery
  The required amounts of analgesics (morphine/paracetamol) during hospital stay; The use of analgesics three months, six months and one year after cardiac surgery, measured with questionnaires;
Genetic variances | Blood sample at time of surgery
  Genetic variances involved in pain sensitivity (e.g. GTP-cyclohydrolase 1 (GCH-1), WDFY4, Zinc Finger gene Family (ZNF), Melanocortin 1 Receptor (MC1R)) and pharmacokinetics and pharmacodynamics of opiates (e.g. glucuronosyl transferase (UGT), Multidrug Resistance-associated Protein (MRP), mu-opioid receptor gene 1 (OPRM1), Catechol-O-methyltransferase (COMT))
Total medical costs and productivity costs during one year, including costs of hospitalization days (ICU and non-ICU) and costs of medications | 1 year after surgery
Mean pain NRS (Numerical Rating Scale) | 3-5 days during hospitalization
  Mean NRS score during intensive care unit (ICU) stay and hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: CAJ Knibbe, Prof. Dr., Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands

REFERENCES:
- [Derived] de Hoogd S, Valkenburg AJ, van Dongen EPA, Daeter EJ, van Rosmalen J, Dahan A, Tibboel D, Knibbe CAJ. Short- and long-term impact of remifentanil on thermal detection and pain thresholds after cardiac surgery: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jan;36(1):32-39. doi: 10.1097/EJA.0000000000000887. PMID 30211725
- [Derived] de Hoogd S, Ahlers SJGM, van Dongen EPA, van de Garde EMW, Daeter EJ, Dahan A, Tibboel D, Knibbe CAJ. Randomized Controlled Trial on the Influence of Intraoperative Remifentanil versus Fentanyl on Acute and Chronic Pain after Cardiac Surgery. Pain Pract. 2018 Apr;18(4):443-451. doi: 10.1111/papr.12615. Epub 2017 Sep 28. PMID 28741894
- [Derived] de Hoogd S, Ahlers SJ, van Dongen EP, Tibboel D, Dahan A, Knibbe CA. Remifentanil versus fentanyl during cardiac surgery on the incidence of chronic thoracic pain (REFLECT): study protocol for a randomized controlled trial. Trials. 2014 Nov 27;15:466. doi: 10.1186/1745-6215-15-466. PMID 25429720
- See also: Study protocol — http://www.ncbi.nlm.nih.gov/pubmed/25429720